CLINICAL TRIAL: NCT03761277
Title: Embrace TDD: Prospective, Multi-Center, Post Market Study to Evaluate Intrathecal (IT) Morphine as an Alternative to Systemic Opioids for the Treatment of Chronic, Intractable, Non-Malignant Primary Back Pain With or Without Leg Pain
Brief Title: Embrace TDD: Post-Market Study to Evaluate Intrathecal Morphine as an Alternative to Systemic Opioids for Chronic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT18026
Record Dates: First submitted 2018-11-15; First posted 2018-12-03 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Chronic Non-malignant Pain; Chronic Pain; Pain, Back; Pain, Leg
Keywords: Pain; Intrathecal; Targeted Drug Delivery (TDD); Non-Malignant Pain; Systemic Opioids; Opioid Weaning; Pain Pump; Drug Pump; Medtronic Pump
MeSH Terms: conditions — Chronic Pain; Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intrathecal Therapy (Other): Enrolled subjects who successfully wean from all systemic opioids and have a successful intrathecal trial, proceed to the intervention phase. This includes implantation with a SynchroMed™ II infusion system in the intrathecal space for targeted drug delivery of preservative-free morphine sulfate (PFMS).
  Interventions: Device: Medtronic SynchroMed™ II infusion system; Drug: Preservative-free morphine sulfate (PFMS)

INTERVENTIONS:
Device: Medtronic SynchroMed™ II infusion system — Implanted infusion system consisting of a pump and catheter, as well as external components of a clinician programmer, refill and catheter access port kits, and the Personal Therapy Manager (myPTM™).
Drug: Preservative-free morphine sulfate (PFMS) — The pharmacological agent used in the pump for this study is limited to a preservative-free morphine sulfate (PFMS).

SUMMARY:
This is a prospective, multi-center, post market study to evaluate Intrathecal (IT) preservative-free morphine sulfate (PFMS) using the SynchroMed™ II infusion system as an alternative to systemic opioids for the treatment of chronic, intractable, non-malignant primary back pain with or without leg pain.

DETAILED DESCRIPTION:
Subjects will be assessed for pain control and opioid-related side effects following a route of delivery change from systemic opioids to IT morphine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide a signed and dated (Medtronic and Institutional Review Board (IRB) approved) Informed Consent Form (ICF) and Health Insurance Portability and Accountability Act (HIPAA) Authorization Form prior to any study procedures being performed
2. A candidate per labeling for the Intrathecal Drug Delivery System (IDDS)
3. A diagnosis of chronic, intractable, non-malignant primary back pain with or without leg pain, treatable with the IDDS
4. Current daily systemic opioid dose of >0 and ≤ 120 Morphine Milligram Equivalents (MME)
5. A Visual Analogue Scale (VAS) of ≥50 mm for pain intensity at the Baseline Visit and/or a Numerical Opioid Side Effect (NOSE) Assessment Tool ≥40 for intolerable side effects at the Baseline Visit
6. Psychological evaluation or investigator assessment of patient psychological suitability for study participation
7. Has an MRI or CT prior to enrollment verifying patent spinal canal and no clinical change in status since last imaging
8. At least 18 years old at time of enrollment
9. Willing and able to attend visits and comply with the study protocol
10. Male or non-pregnant, non-lactating female. Females must be post-menopausal or surgically sterile; or be utilizing a medically acceptable form of birth control (i.e. a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide) for the duration of the study

Exclusion Criteria:

1. Previously trialed or implanted with an IDDS
2. Concomitant stimulation device implanted for the treatment of pain
3. Any ongoing health condition that would be expected to interfere with pain and/or quality of life ratings (i.e. active malignancy, other painful conditions not treatable with IT therapy, etc.)
4. Psychological or other health conditions, financial and/or legal concerns that would interfere with the subject's ability to fulfill the requirements of the protocol as per the investigator's discretion
5. Substance Use Disorder (SUD) within the last 2 years or current Medication Assisted Treatment (MAT) for substance use disorder
6. Currently using cannabinoids or illicit drugs
7. History of allergy or significant adverse reaction to morphine per investigator discretion
8. Currently participating or plans to participate in another investigational study unless written approval is provided by Medtronic Study Team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Neuroversion, Anchorage, Alaska
  - Coastal Pain and Spinal Diagnostics, Carlsbad, California
  - Napa Valley Orthopaedic Medical Group, Napa, California
  - Florida Pain Institute, Merritt Island, Florida
  - Regional Brain & Spine, LLC, Cape Girardeau, Missouri
  - Christian Hospital Pain Management, St Louis, Missouri
  - Comprehensive and Interventional Pain Management, Henderson, Nevada
  - The Pain Management Center, Voorhees Township, New Jersey
  - Premier Pain Treatment Institute, Mount Orab, Ohio
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - Moss Rehabilitation-Einstein Healthcare Network, Elkins Park, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Precision Spine Care, Tyler, Texas
  - University of Virginia Pain Management Center, Charlottesville, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Northwest Pain Care, Inc., Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith TJ, Staats PS, Deer T, Stearns LJ, Rauck RL, Boortz-Marx RL, Buchser E, Catala E, Bryce DA, Coyne PJ, Pool GE; Implantable Drug Delivery Systems Study Group. Randomized clinical trial of an implantable drug delivery system compared with comprehensive medical management for refractory cancer pain: impact on pain, drug-related toxicity, and survival. J Clin Oncol. 2002 Oct 1;20(19):4040-9. doi: 10.1200/JCO.2002.02.118. PMID 12351602
- [Background] Hamza M, Doleys D, Wells M, Weisbein J, Hoff J, Martin M, Soteropoulos C, Barreto J, Deschner S, Ketchum J. Prospective study of 3-year follow-up of low-dose intrathecal opioids in the management of chronic nonmalignant pain. Pain Med. 2012 Oct;13(10):1304-13. doi: 10.1111/j.1526-4637.2012.01451.x. Epub 2012 Jul 30. PMID 22845187
- [Background] Grider JS, Etscheidt MA, Harned ME, Lee J, Smith B, Lamar C, Bux A. Trialing and Maintenance Dosing Using a Low-Dose Intrathecal Opioid Method for Chronic Nonmalignant Pain: A Prospective 36-Month Study. Neuromodulation. 2016 Feb;19(2):206-19. doi: 10.1111/ner.12352. Epub 2015 Oct 19. PMID 26477685
- [Background] Hamza M, Doleys DM, Saleh IA, Medvedovsky A, Verdolin MH, Hamza M. A Prospective, Randomized, Single-Blinded, Head-to-Head Long-Term Outcome Study, Comparing Intrathecal (IT) Boluses With Continuous Infusion Trialing Techniques Prior to Implantation of Drug Delivery Systems (DDS) for the Treatment of Severe Intractable Chronic Nonmalignant Pain. Neuromodulation. 2015 Oct;18(7):636-48; discussion 649. doi: 10.1111/ner.12342. Epub 2015 Aug 26. PMID 26307558
- [Background] Wilkes DM, Orillosa SJ, Hustak EC, Williams CG, Doulatram GR, Solanki DR, Garcia EA, Huang LM. Efficacy, Safety, and Feasibility of the Morphine Microdose Method in Community-Based Clinics. Pain Med. 2018 Sep 1;19(9):1782-1789. doi: 10.1093/pm/pnx132. PMID 29016893
- [Background] Grider JS, Harned ME, Etscheidt MA. Patient selection and outcomes using a low-dose intrathecal opioid trialing method for chronic nonmalignant pain. Pain Physician. 2011 Jul-Aug;14(4):343-51. PMID 21785477
- See also: Applicable Product Manual(s) for the SynchroMed II infusion system — http://manuals.medtronic.com/manuals/main/region

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 2019 through 2021 at 16 sites.
Pre-assignment Details: Subjects are considered enrolled at the time the informed consent form is signed. At the Baseline Visit, consented subjects are assessed for eligibility to the study-specific inclusion and exclusion criteria. Subjects who meet all eligibility criteria begin the systemic opioid weaning process prior to initiating the intrathecal drug trial. Subjects with a successful intrathecal trial are eligible for an Intrathecal Drug Delivery System Implant. Non-implanted subjects are exited from the study.
Groups:
- Enrolled Subjects: All consented subjects are considered enrolled in the study. Enrolled subjects do not receive a treatment intervention before Intrathecal Trial. Subjects who met eligibility criteria proceeded to the Intrathecal Trial procedure. The intrathecal drug trial was conducted according to the investigator's standard of care procedures. A successful intrathecal trial was determined by the investigator.
  Subjects with a successful intrathecal trial were eligible for implant of the Intrathecal Drug Delivery System (IDDS).
  Subjects who were implanted with the IDDS were treated via the IDDS with intrathecal preservative-free morphine sulfate (IT PFMS), at a concentration not exceeding 25 mg/mL and 0.9% solution of preservative-free sodium chloride injection (USP) for dilution. IT PFMS initiation and subsequent dosing adjustments were determined based on specific patient needs and clinician standard practices, with utilization of the lowest reasonable daily dose of IT PFMS.
Period: Enrollment to Implant
Arm/Group | Enrolled Subjects
Started | 93
Intrathecal Trial | 72
Completed | 52
Not Completed | 41
Not completed — Screen Failure | 17
Not completed — Withdrawal by Subject | 17
Not completed — Physician Decision | 2
Not completed — Site Closure | 3
Not completed — Sponsor Request | 2
Period: Post-Implant to 6 Months
Arm/Group | Enrolled Subjects
Started | 52
Completed | 47
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Site Closure | 2
Period: 6 Months to 12 Months
Arm/Group | Enrolled Subjects
Started | 47
Completed | 19
Not Completed | 28
Not completed — Completed Study under Protocol v3 | 25
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population (n=52) is the subset of enrolled subjects who completed the intrathecal trial and were implanted with an Implantable Drug Delivery System (IDDS). Within the 93 enrolled subjects, 21 exited prior to the intrathecal trial, 20 exited after intrathecal trial and before IDDS implant, and 52 received an IDDS implant.
Groups:
- Targeted Drug Delivery Subjects: All subjects implanted with the Intrathecal Drug Delivery System (IDDS). Subjects were treated via the IDDS with intrathecal preservative-free morphine sulfate (IT PFMS), at a concentration not exceeding 25 mg/mL and 0.9% solution of preservative-free sodium chloride injection (USP) for dilution. IT PFMS initiation and subsequent dosing adjustments were determined based on specific patient needs and clinician standard practices, with the goal to maintain or improve pain control and/or opioid-related side effects (compared to Baseline) with utilization of the lowest reasonable daily dose of IT PFMS. The following IT PFMS dose initiation parameters were recommended: (1) A starting PFMS dose of 0.1 to 0.5 mg/day, or half the effective trial dose, with lower initial PFMS doses considered, and (2) a starting concentration to achieve an estimated pump refill interval of 120 days, but not to exceed 180 days. IT PFMS dose increases or decreases could be made any time throughout the duration of study.
Arm/Group | Targeted Drug Delivery Subjects
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 47
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52
Pain (Visual Analog Scale, VAS, 0-100) [Mean (Standard Deviation); unit: units on a scale] — Pain was assessed with the Visual Analog Scale, ranging from 0-100, where 0 is no pain and 100 is the worst pain.
  units on a scale | 75.5 (13.2)
Numerical Opioid Side Effect Assessment (NOSE, 0-100) [Mean (Standard Deviation); unit: units on a scale] — Opioid-related side effects were assessed using the Numerical Opioid Side Effect Assessment, ranging from 0-100, where 0 is no opioid-related side effects and 100 is the worst opioid-related side effects.
  units on a scale | 21.3 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success at the 6-Month Visit
Description: To characterize the number of subjects with Clinical Success at the 6-Month Visit. Clinical Success is defined as any of the following: 1) Reduced opioid-related side effects (at least a 20% reduction) with equal pain (less than 20% increase or decrease) 2) Reduced pain (at least a 20% reduction) with equal opioid-related side effects (less than 20% increase or decrease) 3) Reduced pain and reduced opioid-related side effects (at least a 20% reduction in both). The number of subjects with Clinical Success at the 6-Month Visit is presented.
Time Frame: Baseline to 6-Month Visit
Population: A subset of the Targeted Drug Delivery Subjects who maintained intrathecal morphine monotherapy (ITMM) and provided outcome data at both the Baseline and 6-Month (6M) Visit. Of the 52 implanted subjects, 47 completed the 6M Visit, and 42 maintained ITMM through the 6M Visit. Four of the subjects who did not maintain ITMM through the 6M Visit changed their intrathecal medication, and one subject was explanted prior to the 6M Visit and completed the 6M Visit post-explant.
Measure: Count of Participants; unit: Participants
Groups:
- Targeted Drug Delivery Subjects: All subjects implanted with the Intrathecal Drug Delivery System (IDDS). Subjects were treated via the IDDS with intrathecal preservative-free morphine sulfate (IT PFMS), at a concentration not exceeding 25 mg/mL and 0.9% solution of preservative-free sodium chloride injection (USP) for dilution. IT PFMS initiation and subsequent dosing adjustments were determined based on specific patient needs and clinician standard practices, with the goal to maintain or improve pain control and/or opioid-related side effects (compared to Baseline) with utilization of the lowest reasonable daily dose of IT PFMS.
Arm/Group | Targeted Drug Delivery Subjects
Number analyzed (Participants) | 42
Participants | 25

2. Secondary Outcome: Visual Analog Scale (VAS) Pain Intensity at the 6-Month Visit
Description: To demonstrate pain intensity scores (Visual Analog Scale, VAS) at the 6-Month Visit is non-inferior to VAS at Baseline, with a non-inferiority margin of 10mm. Pain was assessed using a Visual Analog Scale, ranging from 0-100, where 0 is no pain and 100 is the worst pain. The VAS is a 100mm line, with "No pain" on the left side of the line and "Worst pain imaginable" on the right side of the line. Subjects made a perpendicular mark on the VAS line that best describes their average pain in the last 24 hours. Change in VAS is calculated as 6-Months - Baseline, with a negative change indicating a reduction (i.e., improvement) in pain intensity.
Time Frame: Baseline to 6-Month Visit
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Targeted Drug Delivery Subjects
Number analyzed (Participants) | 42
units on a scale | -15 [-22.7 to -7.1]
Statistical Analysis 1: Comparison: Targeted Drug Delivery Subjects; This analysis was to demonstrate pain intensity scores (VAS) at the 6-Month Visit is non-inferior to VAS at Baseline, i.e., the change in pain intensity is not greater than 0 by more than 10 points from Baseline to the 6-Month Visit; Test type: Non-Inferiority — This analysis was to demonstrate pain intensity scores (VAS) at the 6-Month Visit is non-inferior to VAS at Baseline, i.e., the change in pain intensity is not greater than 0 by more than 10 points from Baseline to the 6-Month Visit, with change calculated as 6-Month - Baseline; p < 0.001, Wilcoxon Signed Rank test; Mean Difference (Final Values) = -15, 97.5% CI 1-sided [upper limit -7.1], Standard Deviation 25.0; Due to non-normality, the non-inferiority test was conducted using a Wilcoxon Signed Rank test, rather than a one-sample t-test. Mean reduction in VAS and the upper 97.5% confidence limit are presented, but the change from baseline was evaluated using non-parametric analysis methods
Statistical Analysis 2: Comparison: Targeted Drug Delivery Subjects; This analysis was to demonstrate pain intensity scores (VAS) at the 6-Month Visit are less than VAS at Baseline, i.e., the reduction in pain intensity is less than 0 from Baseline to the 6-Month Visit; Test type: Superiority — This analysis was to demonstrate pain intensity scores (VAS) at the 6-Month Visit are less than VAS at Baseline, i.e., the reduction in pain intensity is less than 0 from Baseline to the 6-Month Visit, with change calculated as 6-Month - Baseline; p < 0.001, Wilcoxon Signed Rank test; Mean Difference (Final Values) = -15, 95% CI 2-sided [-22.7 to -7.1], Standard Deviation 25.0; Due to non-normality, the superiority test was conducted using a Wilcoxon Signed Rank test, rather than a one-sample t-test. Mean reduction in VAS and 95% confidence interval are presented, but the change from baseline was evaluated using non-parametric analysis methods

3. Secondary Outcome: Numerical Opioid Side Effect (NOSE) Assessment Tool
Description: To characterize the change in opioid-related side effects scores (NOSE) from Baseline to the 6-Month Visit. The Numerical Opioid Side Effect (NOSE) Assessment Tool is a tool to evaluate 10 opioid-related side effects using a 11-point numerical scale. Subjects are asked to evaluate each of the 10 opioid-related side effects on a scale of 0 - 10 with 0 being "not present" and 10 being "as bad as you can imagine". A total sum score can range from 0 - 100, where 0 is no opioid-related side effects and 100 is the worst opioid-related side effects. Change in NOSE is calculated as 6-Months - Baseline, with a negative change indicating a reduction (i.e., improvement) in opioid-related side effects.
Time Frame: Baseline to 6-Month Visit
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Targeted Drug Delivery Subjects
Number analyzed (Participants) | 42
score on a scale | -9.4 [-15.4 to -3.4]

4. Secondary Outcome: Number of Participants With Systemic Opioid Elimination Through the 6-Month Visit
Description: To characterize the number of subjects who eliminate systemic opioids through the 6-Month Visit. Four drug tests for systemic opioid use are administered from intrathecal therapy initiation through the 6-Month Visit. If all of the available drug tests are negative for systemic opioid use, the subject is counted as eliminating systemic opioids through the 6-Month Visit. The number of subjects who eliminated systemic opioids through the 6-Month Visit is presented.
Time Frame: Baseline to 6-Month Visit
Population: The subset of Targeted Drug Delivery Subjects who have a drug test at the 6-Month Visit and no more than 1 missing drug test through the 6-Month Visit. Of the 52 implanted subjects, 47 completed the 6M Visit, 42 maintained ITMM through the 6M Visit, and 41 completed a drug test at the 6-Month and had no more than 1 missing drug test through the 6-Month Visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Drug Delivery Subjects
Number analyzed (Participants) | 41
Participants | 31

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date of subject consent through study exit, up to 12 months following intrathecal therapy initiation after implant of the Intrathecal Drug Delivery System, if applicable.
Description: Any adverse event (AE) meeting the definition of systemic opioid weaning-related, device-related, intrathecal drug-related, and procedure-related, all serious adverse events and deaths (regardless of relatedness) for all subjects from consent to the 12-Month Visit, were collected. Subjects were assessed for adverse events by the investigator at each scheduled and unscheduled study visit.
Groups:
- Enrolled Subjects: All consented subjects are considered enrolled in the study. Enrolled subjects do not receive a treatment intervention before Intrathecal Trial. Subjects who met eligibility criteria proceeded to the Intrathecal Trial procedure. The intrathecal drug trial was conducted according to the investigator's standard of care procedures. A successful intrathecal trial was determined by the investigator.
  Subjects with a successful intrathecal trial were eligible for implant of the Intrathecal Drug Delivery System (IDDS).
  Subjects who were implanted with the IDDS were treated via the IDDS with intrathecal preservative-free morphine sulfate (IT PFMS), at a concentration not exceeding 25 mg/mL and 0.9% solution of preservative-free sodium chloride injection (USP) for dilution. IT PFMS initiation and subsequent dosing adjustments were determined based on specific patient needs and clinician standard practices, with the goal to maintain or improve pain control and/or opioid-related side effects (compared to Baseline) with utilization of the lowest reasonable daily dose of IT PFMS.
Arm/Group | Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 1/93
Serious Adverse Events (participants affected / at risk) | 20/93
Other Adverse Events (participants affected / at risk) | 18/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=93)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Drug withdrawal syndrome (General disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=93)
Urinary retention (Renal and urinary disorders) | 7 (9)
Adverse drug reaction (General disorders) | 9 (14)
Drug withdrawal syndrome (General disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Protocol V3.0 revised the last study visit from the 12-Month Visit to the 6-Month Visit at a point in the study where some subjects, but not all, had already progressed beyond the 6-Month Visit. Thus, subjects consented under Protocol V3.0 may complete the study without completing the 12-Month Visit. This protocol revision did not impact the Primary and Secondary endpoints, which are evaluated at 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No manuscripts, abstracts, or case reports that jeopardize the primary publication will be submitted prior to the submission of the primary publication. It is required that all publications undergo review at Medtronic for confidential information and technical accuracy prior to publication.

DOCUMENTS (2):
  • Study Protocol (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT03761277/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT03761277/SAP_001.pdf